CLINICAL TRIAL: NCT02829671
Title: Study of Loneliness as Predictive Factor for Suicidal Behavior
Brief Title: Loneliness and Occurrence of Suicide Attempts and Suicidal Ideas
Acronym: SOLSTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF 9702; 2016- -A00276-45 (Other: FRANCE: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Major Depressive Disorders
Keywords: Loneliness; Suicidal behavior; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with major depressive disorders (Other)
  Interventions: Other: Clinical and biological assessment

INTERVENTIONS:
Other: Clinical and biological assessment — Blood sample, clinical assessment with questionnaires

SUMMARY:
Suicide is a major health problem that causes annually a million death worldwide. Loneliness is known to be associated with suicidal ideation in minors and to be related with suicidal risk in elderly people. However little is known about this association in a middle-aged population. Loneliness is a modifiable factor with suitable psychotherapeutic measures, it is essential to improve the scientific and medical knowledge about the link between this feeling and suicide risk in a population of depressed patients in middle age.

The main objective is the study of the relationship between loneliness and the occurrence of suicidal behavior (SB) in major depressed adult population over 12 months.

The secondary objectives are:

* Identification of risk factors (clinical, neuropsychological and biological) of the occurrence of SB within a clinical population and their interaction;
* Identification of predictive factors (clinical, neuropsychological, biological) therapeutic response to antidepressant in the context of depression.

DETAILED DESCRIPTION:
This project is based on clinical, neuropsychological and biological data routinely collected in the Department of Emergency Psychiatry and Post Acute Care. This is a one year follow-up prospective study.

Over three years, 600 depressed patients will be recruited.

* First visit (inclusion): clinical, biological and neuropsychological assessment
* Follow up visits (3, 6 and 12 months): clinical assessment only

ELIGIBILITY:
Inclusion criteria:

Main diagnosis of major depressive disorder according to Diagnostic and Statistical Manual of Mental DisordersIV (DSM IV) Having signed informed consent Able to understand nature, aims, and methodology oh the study

Exclusion criteria:

Participation in another clinical trial Patient on protective measures (guardianship or trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
frequency of suicide attempts at one year | At 12 months
  frequency of suicide attempts during the 12 months follow-up depending on the intensity of the feeling of loneliness evaluated by the loneliness scale of the University of Laval (ESUL)

SECONDARY OUTCOMES:
frequency of suicide attempts during the follow up | At 3 and 6 months
  frequency of suicide attempts during the follow up
comorbid psychiatric disorders of Axis I | At the inclusion, 3, 6, and 12 months
  comorbid psychiatric disorders of Axis I assessed by the Mini International Neuropsychiatric Interview (MINI)
intensity of the depression | At the inclusion, 3, 6, and 12 months
  intensity of the depression assessed by the physician with the Inventory of Depressive Symptomatology, clinician rating (IDSC-30) and with the Montgomery-Asberg depression rating scale (MADRS) and assessed by the patient with the Beck Depression Inventory (BDI) scale.
intensity of suicidal ideation | At the inclusion, 3, 6, and 12 months
  intensity of suicidal ideation assessed by visual analogic scale
features of suicidal behavior | At the inclusion, 3, 6, and 12 months
  Features of SB (number and methods of suicide attempts, nature of the precipitating factor, motivation, lethality, level of impulsiveness or premeditation) by the Columbia-Suicide Severity Rating Scale (CSSRS), the Risk Rescue Rating Scale (RRRS) and the Suicidal Intent Scales (SIS).
personal history of childhood abuse | At the inclusion, 3, 6, and 12 months
  personal history of childhood abuse assessed by the Childhood Trauma Questionnaire
intensity of psychological pain | At the inclusion, 3, 6, and 12 months
  intensity of psychological pain assessed by visual analogic scale
inflammatory markers | At the inclusion, 3, 6, and 12 months
  level of C protein reactive in a blood sample collected at inclusion
thyroid function | At the inclusion
  levels of thyroid-stimulating hormone (TSH), triiodothyronine(T3), and thyroxine(T4) in a blood sample collected at inclusion
lipid profile | At the inclusion
  level of cholesterol, triglycerides, phospholipids in a blood sample collected at inclusion

IPD SHARING:
Plan to Share IPD: No